CLINICAL TRIAL: NCT04759729
Title: The Effect of Probiotics and Vitamin D Supplementation on Sport Performance and Intestinal Barrier Function in Trained Male Mixed-martial Arts Athletes
Brief Title: The Effect of Probiotics and Vitamin D Supplementation on Sport Performance in MMA Athletes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Gdansk (Other)
Collaborators: Gdansk University of Physical Education and Sport (Other); Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MMA29012021
Record Dates: First submitted 2021-02-07; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Gut Microbiome; Sport Performance
Keywords: microbiota; sport performance; mixed-martial arts; microbiome; vitamin D
MeSH Terms: interventions — Probiotics; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO+D group (Experimental): Participants will receive probiotic as well as vitamin D supplementation.
  Interventions: Combination Product: Probiotic and vitamin D
- PL+D group (Experimental): Participants will receive placebo instead of probiotics and vitamin D supplementation.
  Interventions: Dietary Supplement: placebo and vitamin D

INTERVENTIONS:
Combination Product: Probiotic and vitamin D — Participants enrolled to PRO + D group will receive probiotics and vitamin D supplements as a intervention product.
  Participants enrolled to probiotic group will receive probiotics as well as vitamin D supplements.
  Arms: PRO+D group
Dietary Supplement: placebo and vitamin D — Participants enrolled to PL+D group will receive vitamin D. Additionally they will get placebo instead of probiotics.
  Arms: PL+D group

SUMMARY:
The probiotics supplementation seems to be safety way to optimize the intestinal microbiota composition and thus modulate the immune system and reduce oxidative stress. Moreover it may enhance muscle protein synthesis, mitochondrial biogenesis and function, as well as muscle glycogen storage. Probiotics intake via reduce inflammatory markers and reactive oxygen species production may attenuate macromolecules damage and have some beneficial effect on aerobic and anaerobic performance. The combined probiotics and vitamin D supplementation may enhance this effect. The synergistic intestinal microbiota and vitamin D interaction towards muscle protein synthesis and mitochondrial function improvement may be manifested by mTOR and FOXO signaling influence on oxidative stress as well as immunological functions modulation. In the study investigators will assess if multistrain probiotic mixture in conjunction with vitamin D may have beneficial effect on sport performance among trained male mixed-martial arts athletes. The study protocol is designed as a randomized double-blind placebo-controlled clinical trial. Researchers are going to evaluate changes in the gut, including microbiome composition and epithelial permeability; differences in the blood parameters as well as direct influence on sport performance, expressed by anaerobic and aerobic fitness capacity. Researchers will provide an evidences, having both theoretical as well as practical aspect.

DETAILED DESCRIPTION:
The study is designed as a randomized double-blind placebo-controlled clinical trial with 4-week probiotics and vitamin D intervention period. The study is conducted between December 2020 and March 2021, at the Medical University of Gdańsk, Department of Bioenergetics and Physiology of Exercise (Gdańsk, Poland) . Researchers will enrol 25 trained, male mixed-martial arts athletes. Enrolled athletes will be randomly assigned to receive probiotic (PRO) or matching placebo (PL) in a 1:1 ratio, using Excel random number generator, following the rule of the random and blindness.

The study product is a vitamin D ,,Juvit d3" and probiotic mixture ,,Sanprobi Active & Sport", containing 2,5 x 109 CFU/g per capsule (≥500 million CFU in one capsule) of five strains of lactic acid bacteria (Bifidobacterium lactis W51, Lactobacillus brevis W63, Lactobacillus acidophilus W22, Bifidobacterium bifidum W23 and Lactococcus lactis W5); maize starch, maltodextrin, plant proteins and hydroxypropyl ethylcellulose tablets' coating. Identical-looking placebo capsules containing 40 mg of maltodextrin and plants proteins will be used for cartel. Each pack of probiotic or placebo contain 40 capsules. All athletes will receive a bottle of Juvit d3 as well as three identical-looking packings of probiotics or placebo, depending on the random allocation, at the baseline visit. Participants will be informed to take 4 capsules with meals and 3500 iu of vitamin d daily.

At baseline visit, all subjects will receive the study product as well as diary of supplements and dietary intake and training diary. Both PRE and POST visit will be splitted in two days in order to reliable and appropriate performance of all procedures. The time window between these splitted visit is 3-5 days. Participants will report to the Medical University of Gdańsk at the beginning (PRE) and the end (POST) of the 4-week intervention period. During both visits athletes will complete an assessment of body composition, food frequency questionnaire (FFQ), cardio-respiratory fitness evaluation and will provide fecal samples. Furthermore, the blood samples will be drawn before and after sport tests, to assess selected markers of inflammatory as well as muscle damage state and lactate utilization level. The last one blood collection will be perform after 24 hours of anaerobic sport test. Participant will be instructed to continue their training programme. Athletes will be obligated to perform at least 5 endurance workouts per week to keep the competitive character of the study.

The body composition analysis will be evaluated to detect potential changes within body fat mass and fat free mass. The level of each tissue will be compared to intestinal bacteria content. Investigators will try to explain if gut microbiome composition may affect body composition and which bacterial phyla are responsible for possible for this potential changes. This target will be obtain through multi-frequency bioelectrical impedance analysis (BIA).

Aerobic fitness capacity will be assess through bicycle ergometer ER900 Jaeger using the wasserman protocol. The test will be preceded by a 5-minute warm-up with a load of 100 W, followed by a 5-minute rest. The test will start at a load of 125 W and a frequency of 60 ± 5 RPM / min, the load will be increased every 1 minutes by 25 W. The test will be conducted until the maximum individual exercise load is reached, i.e. the inability to continue the exercise while maintaining the specified frequency or lack of increase oxygen uptake. During examination investigators will monitor the amount of oxygen uptake and carbon dioxide exhaled, minute lung ventilation as well as heart rate. The aerobic test will be conducted 3-5 days before anaerobic assessment as part of PRE and POST visits.

Anaerobic fitness assessment will be obtained by the Wingate Anaerobic Test (WAnT) using cycloergometer MCE_v_5.1. Before the examination, the saddle will be individually adjusted, then the athletes will perform a 5-minute warm-up at 50 W load and a frequency of 60 RPM / min, with two 10-second accelerations in 3 and 4 minutes. After the warm-up, there will be a 3-minute rest. The load will be adjusted individually and will amount to 7.5% of the athlete's body weight. At the "start" command, the athlete will performing a 30-second sprint in a sitting position, trying to achieve peak power as quickly as possible and maintain it throughout the duration of the effort. After the test, there will be an active 2-minute break. The test will be carried out 3 times. The WAnT assesses the maximum, minimum and average power, time to reach maximum power and relative power drop.

The blood samples will be collected during Wingate tests at the two points time: PRE and POST intervention, at the same conditions. Blood samples from the arm vein will be drawn by a specialist nurse into two appropriate standardized tubes containing respectively K2EDTA and clotting activator. Each time up to 4 ml of blood will be collected. Blood samples will be taken indirectly before the start of exercise tests, 30 minutes after the end of the tests and 24 hours after the end of the tests. The blood will then be centrifuged at 3000 x g to separate serum and plasma. The material will be placed into separately labeled microcentrifuge tubes and stored at -80 ° C for later determinations. All analysis will be performed at the end of the study at Medical University in Gdańsk.

The collected venous blood samples will be subjected to analysis at the Medical University of Gdańsk. Researchers will assess the level of serum pro-inflammatory cytokines (IL-6 and TNF-α) as well as anti-inflammatory cytokines (L-2 and IL-15) using a commercially available enzyme-linked immunosorbent assay (ELISA) kits. To evaluate the plasma level of muscle damage investigators will determinate the activity of creatine kinase (CK) through kinetic method, using the commercially available kit.

Capillary blood samples will be taken each time, Wingate tests are performed, by a specialized nurse, in an amount of 100 µL, into a sterile graduated microcapillary. The measurements will be performed on fingertip capillary blood. The blood will then be transferred to a micro-centrifuge tube containing 500 µl 0.6 mol perchloric acid, centrifuged and stored at -20 degrees C until the determination is carried out. Capillary blood will be collected before exercise testing and in 2-3, 15, 30 and 60 minutes after test. Collected capillary blood samples will undergo analysis at the Medical University of Gdańsk. The purpose of the analysis will be to determine the level of lactate in the samples taken. Determination of lactate level will be performed using colorimetric kinetic method, based on reaction speed.

The subjects will provide a fecal sample indirectly before and after the intervention period. The material will be collected by participants into a special standardized container. A stool sample will be taken twice: before testing, and in the end of the intervention. Stool samples will be immediately frozen and stored at -80 degrees Celsius, then in the same conditions transported to the assessment by independent laboratory. Collected fecal samples will be subjected to quantitative and qualitative content of the intestinal microbiota with using the new generation sequencing method. Selected hypervariable regions of the 16SrRNA gene will be analyzed. The composition of the microbiome will be characterized primarily by alpha and beta diversity. Diversity of microbial communities in one sample (alpha) will be measured using several indicators, such as Chao1, ACE, Shannon and inverted Simpson. All indicators will be calculated on the basis of raw NGS data (without any pre-processing, e.g. removal of rare species) and compared between the test and control group using a standard statistical test depending on the distribution of variables. Diversity of microbial communities between samples (beta) will be measured using the difference indicator (Bray-Curtis) and distance metrics (UniFrac weighted - a phylogenesis-based metric). Similarity indicators will be calculated for all sample pairs and stored in dissimilarity matrices. Bray-Curtis will perform permutation multivariate analysis of variance (PERMANOVA) and weighted UniFrac difference matrices to assess differences at the group level. Beta diversity analysis will be preceded by supervised and unattended pre-processing of data, such as the removal of rare species and transformation of numbers using the median sequencing depth as a scaling factor. Collected fecal samples will be analyzed in the context of the presence of intestinal permeability parameters such as calprotectin, zonulin and IFABP as well as bacterial metabolism products such as short chain fatty acids (SCFA).

All obtained data will be analysed using the statistic program Statistica 13. To statistical analysis will be included only full data, from subjects who complete all intervention period as well as all study procedures. Data will be previously checked for normality using Shapiro-Wilk W-test. In the case of data' abnormal distributed, their natural logarithms will be used. Researchers will usual descriptive statistics for background information as well as to examine the trends in the analysed parameters with mean values of 95% confidence interval. Depending on the normality of the underlying data, parametric or non-parametric tests will be carried out. The statistical significance is set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* male gender
* signed informed consent
* minimum 3 years of mixed martial arts training practice
* realization of minimum 5 workouts weekly
* participation in 2 competitions at least

Exclusion Criteria:

* age below 18
* female gender
* lack of signed informed consent
* antibiotic therapy during last 3 months
* diagnosed inflammatory bowel disease
* chronic musculoskeletal injuries within last 6 months
* heart failure or defects

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of changes in gut microbiome composition caused by intervention. | Participants will be obligated to deliver a stool samples at the baseline and follow up visit. The outcome measure will be assessed up to 9 months
  Collected stool samples will be assessed with new generation sequencing method. Selected hypervariable regions of the 16SrRNA gene will be analyzed. The composition of the microbiome will be characterized primarily by alpha and beta diversity. Diversity of microbial communities in one sample (alpha) will be measured using several indicators, such as Chao1, ACE, Shannon and inverted Simpson. During the analysis investigators will assess presence of short-chain fatty acid.
Evaluation of changes in the gut on epithelial permeability | Participants will be obligated to deliver a stool samples at the baseline and follow up visit. The outcome measure will be assessed up to 9 months
  Collected stool samples will be assessed in the context intestine barrier permeability as zonulin, calprotectin and FABP.
Assessment of changes in body composition c.used by intervention, | The measurement will be perform in the morning, at baseline and follow up visit (before sport tests, before breakfast). The outcome measure will be assessed up to 1 month.
  The body composition analysis will be evaluated to detect potential changes within body fat mass and fat free mass. The level of each tissue will be compared to intestinal bacteria content. Investigators will try to explain if gut microbiome composition and vitamin D may affect body composition and which bacterial phyla are responsible for possible for this potential changes. This target will be obtain through multi-frequency bioelectrical impedance anap visit (before sport tests, before breakfast). The outcome measure will be assessed up to 1 month (BIA)
The effect of probiotics and vitamin D supplementation on inflammatory state- the evaluation on changes between baseline and follow up visit. | The arm vein blood will be collected at baseline as well as follow up visit at three time points - before breakfast and sport tests, 35 minutes after anaerobic tests and 24 hours after Wingate test. The outcome measure will be assessed up to 6 months
  The collected venous blood samples will be subjected to analysis at the Medical The effect of probiotics and vitamin D supplementation on inflammatory state - the evaluation on changes between baseline and follow up visit. The outcome measure will be assessed up to 6 monthsUniversity of Gdańsk. Investigators will assess the level of serum pro-inflammatory cytokines (IL-6 and TNF-α) as well as anti-inflammatory cytokines (L-2 and IL-15) using a commercially available enzyme-linked immunosorbent assay (ELISA) kits.
The effect of probiotics and vitamin D supplementation on muscle damage - the evaluation on changes between baseline and follow up visit. | The arm vein blood will be collected at baseline visit at three time points - before breakfast and sport tests, 35 minutes after anaerobic tests and 24 hours after Wingate test. The outcome measure will be assessed up to 6 months .
  The collected venous blood samples will be subjected to analysis at the Medical University of Gdańsk.Investigators will assess changes in creatine kinase level through kinetic method, using the commercially available kit.
Effect of probiotics and vitamin D supplementation on aerobic sport performance - evaluation of changes | Aerobic test will be perform 3-5 days before/after anaerobic test. The outcome measure will be assessed up to 3 months.
  To assess an effect on aerobic sport performance investigators will perform aerobic (cardio-pulmonary exercise test) as well as anaerobic test (triple Wingate test) using cycloergometer. Additionally the capillary blood will be collected to assess the level of lactate concentration as well as rate of lactate utilization.
Effect of probiotics and vitamin D supplementation on anaerobic sport performance - evaluation of changes | The Wingate test will be perform at baseline and follow up visit. The outcome measure will be assessed up to 3 months .
  To assess an effect on sport performance investigators will perform anaerobic triple Wingate test using cycloergometer.
Effect of probiotics and vitamin D supplementation on lactate utilization - evaluation of changes | Capillary blood will be collected in 5 time points, directly before Wingate test, 3, 15, 30 and 60 minutes after test.The outcome measure will be assessed up to 3 months
  The capillary blood will be collected to assess the level of lactate concentration as well as rate of lactate utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna KP Przewłócka, MSc, Principal Investigator — Medical University of Gdańsk, Gdańsk, Poland
Locations (1):
- Medical University of Gdańsk, Gdansk, Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No